CLINICAL TRIAL: NCT02349555
Title: An Open-Label Single-Center Study to Determine Safety and Effects of Novel Nutritional Blend on Inflammatory Balance Markers and Metabolic Parameters
Brief Title: Nutritional Supplement Impact on Metabolic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: Texas Diabetes & Endocrinology, P.A. (Other); Utah State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14-PHX-0001
Record Dates: First submitted 2015-01-15; First posted 2015-01-29 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Other Endocrine/Nutritional/Metabolic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutritional Supplement Blend (Experimental): The nutritional supplement contains a proprietary blend consisting of 15 unique nutritional ingredients.
  Interventions: Dietary Supplement: Nutritional Supplement Blend

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement Blend — It is to be taken orally at a dose of 4 capsules per day, 2 capsules with breakfast and 2 capsules with dinner.

SUMMARY:
This open label study seeks to study the effects of a nutritional supplement on inflammatory markers, metabolic parameters, and safety in subjects compared to baseline after taking supplement for 2 and 4 months.

DETAILED DESCRIPTION:
Primary endpoint will be to determine if nutritional supplement decreases the metabolic parameter of triglycerides. Numerous studies have demonstrated the efficacy of fish oil on reducing triglycerides in subjects taking fish oil at similar doses provided in our product (see references).

Additional metabolic parameters will be measured as secondary endpoints, including abdominal obesity, HDL cholesterol, blood pressure, fasting glucose, haemoglobin A1c, skin glycation (AGEs), pulse wave velocity, skin carotenoids, serum 25(OH)D concentrations, weight, and LDL density, particle size and number. The novel nutritional supplement contains many nutrients that have been shown to improve metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Subject male or female between the ages of 30-70 at the time of informed consent.
2. Fasting Blood Glucose between 90 and 125mg/dL in the serum and 2 additional parameters at screening:

   * Abdominal obesity defined by >102 cm (>40in) waist circumference in men and >88cm (>35in) waist circumference in women, or
   * Triglycerides ≥ 150mg/dL, or
   * HDL cholesterol <40 mg/dL in men and <50 mg/dL in women
3. Hemoglobin A1C less than 6.5% at screening
4. BMI >27kg/m2
5. Blood Pressure <150/90 mm Hg
6. Subject is willing and able to comply with study restrictions, procedures, and assessments.
7. Subject is able to swallow product without difficulty.
8. Subject is willing to fast for 8h prior to blood draw at screening, baseline, 2 month, and 4 month visits.
9. Subject is willing to maintain usual diet and physical activity for the duration of the study.
10. Eats 1 or fewer servings of fatty fish per week (e.g. salmon, tuna, mackerel, herring, anchovies, etc.)
11. Subject is willing to take the study multi-vitamin/mineral supplement for 30 days prior to starting investigational product and during the 4 month intake of investigational product.
12. Use of effective method of contraception by females of childbearing potential 30-days before the screening visit and agree to continue to practice that acceptable method of contraception for the duration of her participation in the study. Acceptable methods of contraception include oral, injectable, or implantable contraceptives; intrauterine devices, diaphragm plus spermicide; abstinence (must agree to use double-barrier method if they become sexually active), transdermal patch, or any double barrier method including a vasectomized sexual partner. Women who have had a hysterectomy (partial or total) or tubal ligation at least 6 months prior to Visit 1 or who have been post-menopausal for at least 1 year prior to Visit 1 are not considered to be of childbearing potential.

Exclusion Criteria:

1. Subject has a known allergy or intolerance to any of the ingredients contained in the nutritional supplement.
2. Subject currently uses nicotine or has not quit using for at least 1 year.
3. Subject is taking an unapproved medication or has not been on a stable dose, for at least 8 weeks, of approved medication.
4. Subject who has undergone any type of surgery on their intestines that would interfere with product absorption, in the opinion of the investigator.
5. Subject is not willing to stop taking dietary/nutritional supplements for duration of study.
6. Subject is taking any dietary/nutritional supplements, not provided by the sponsor, within 30 days prior to investigational product administration.
7. Abnormalities in screening laboratory samples that the investigator would consider unstable/unsafe.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Serum Triglycerides at 2 months and 4 months | Baseline, 2 months, 4 months

SECONDARY OUTCOMES:
Change from Baseline in Abdominal Obesity at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in HDL cholesterol at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Fasting glucose at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Total cholesterol at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in LDL density, particle size, and number at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Hemoglobin A1c at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Skin glycation (AGEs) at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Pulse wave velocity measurements at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Erythrocyte sedimentation rate at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Cytokine and additional markers at 2 months and 4 months | Baseline, 2 months, 4 months
  TNF-α, TNF Receptors 60 and 80, IL-1β, IL-6, IL-1, IL-2, ICAM-1, hsCRP, IL-10, sVCAM-1, insulin, leptin, and adiponectin
Change from Baseline in Serum 25(OH)D concentrations at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Skin carotenoids at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Weight at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Red blood cell fatty acid profile at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Chemistry panel at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Thyroid panel at 2 months and 4 months | Baseline, 2 months, 4 months
Change from Baseline in Vital signs at 2 months and 4 months | Baseline, 2 months, 4 months
  Heart Rate and Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blevins, MD, Principal Investigator — Founder; Michael Lefevre, PhD, Principal Investigator — Scientific Director
Locations (2):
- United States (2):
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Utah State University, Logan, Utah

REFERENCES:
- [Background] Tavazzi L, Maggioni AP, Marchioli R, Barlera S, Franzosi MG, Latini R, Lucci D, Nicolosi GL, Porcu M, Tognoni G; Gissi-HF Investigators. Effect of n-3 polyunsaturated fatty acids in patients with chronic heart failure (the GISSI-HF trial): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Oct 4;372(9645):1223-30. doi: 10.1016/S0140-6736(08)61239-8. Epub 2008 Aug 29. PMID 18757090
- [Background] Earnest CP, Kupper JS, Thompson AM, Guo W, Church T. Complementary effects of multivitamin and omega-3 fatty acid supplementation on indices of cardiovascular health in individuals with elevated homocysteine. Int J Vitam Nutr Res. 2012 Feb;82(1):41-52. doi: 10.1024/0300-9831/a000093. PMID 22811376
- [Background] Ebrahimi M, Ghayour-Mobarhan M, Rezaiean S, Hoseini M, Parizade SM, Farhoudi F, Hosseininezhad SJ, Tavallaei S, Vejdani A, Azimi-Nezhad M, Shakeri MT, Rad MA, Mobarra N, Kazemi-Bajestani SM, Ferns GA. Omega-3 fatty acid supplements improve the cardiovascular risk profile of subjects with metabolic syndrome, including markers of inflammation and auto-immunity. Acta Cardiol. 2009 Jun;64(3):321-7. doi: 10.2143/AC.64.3.2038016. PMID 19593941
- [Background] Hill AM, Buckley JD, Murphy KJ, Howe PR. Combining fish-oil supplements with regular aerobic exercise improves body composition and cardiovascular disease risk factors. Am J Clin Nutr. 2007 May;85(5):1267-74. doi: 10.1093/ajcn/85.5.1267. PMID 17490962
- [Background] Vanschoonbeek K, Feijge MA, Paquay M, Rosing J, Saris W, Kluft C, Giesen PL, de Maat MP, Heemskerk JW. Variable hypocoagulant effect of fish oil intake in humans: modulation of fibrinogen level and thrombin generation. Arterioscler Thromb Vasc Biol. 2004 Sep;24(9):1734-40. doi: 10.1161/01.ATV.0000137119.28893.0b. Epub 2004 Jun 24. PMID 15217806
- [Background] Garg ML, Blake RJ, Clayton E, Munro IA, Macdonald-Wicks L, Singh H, Moughan PJ. Consumption of an n-3 polyunsaturated fatty acid-enriched dip modulates plasma lipid profile in subjects with diabetes type II. Eur J Clin Nutr. 2007 Nov;61(11):1312-7. doi: 10.1038/sj.ejcn.1602650. Epub 2007 Feb 7. PMID 17299483